CLINICAL TRIAL: NCT01492413
Title: Impact of an Online Behavioral Weight Loss Program Provided With or Without a Fortified Diet Beverage
Brief Title: Impact of an Online Behavioral Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Beverage Institute. (Unknown); Temple University (Other); MRC Human Nutrition Research (Other Government); National Development and Research Institutes, Inc. (Other)
Responsible Party: Principal Investigator, John P. Foreyt, Professor, Department of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BI-001
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Online basic lifestyle counseling (OBLI) (Experimental): Subjects receive one online informational class.
  Interventions: Behavioral: online lifestyle counseling and a fortified diet beverage
- Online lifestyle counseling (OLC) (Experimental): Subjects receive 12 weekly online classes with a focus on behavior modification for weight loss.
  Interventions: Behavioral: online lifestyle counseling and a fortified diet beverage
- OBLI intervention plus a fortified diet beverage (BEV) (Experimental): Subjects receive online basic lifestyle information (OBLI) plus a fortified diet beverage.
  Interventions: Behavioral: online lifestyle counseling and a fortified diet beverage
- OLC plus fortified diet beverage (BEV) (Experimental): Subjects receive OLC plus diet beverage (BEV).
  Interventions: Behavioral: online lifestyle counseling and a fortified diet beverage

INTERVENTIONS:
Behavioral: online lifestyle counseling and a fortified diet beverage — The fortified diet beverage contains green tea extract (total catechin 167 mg), soluble dextrin fiber (10 g), and caffeine (100 mg).

SUMMARY:
This study was designed to test the impact of a 12-week online behavioral modification program for weight loss, with or without a fortified beverage. Subjects are randomized to four conditions: 1) Online Basic Lifestyle Counseling (OBLI); 2) Online Lifestyle Counseling (OLC); 3) OBLI plus a beverage (BEV); 4) OLC + BEV. The three hypotheses were: 1)after 12 weeks, individuals in the OLC condition would lose more weight than those in OBLI; 2) after 12 weeks, the OLC + BEV condition would lose more weight than the OLC condition; and 3) after 12 weeks, the OBLI + BEV condition would lose more weight than the OBLI condition.

DETAILED DESCRIPTION:
This study tests the impact of an innovative combination of a fortified beverage (a diet cola containing green tea extract, soluble dextrin fiber, and caffeine) and an online support weight loss program in a multi-center randomized clinical trial. The study compares the impact of all combinations of the beverage and the online behavioral modification treatment program over 12 weeks at three treatment center in the US and EU.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) of 25 to 40;
2. age 18 to 65 years;
3. blood pressure less than 140 mmHg systolic and 90 mmHg diastolic;
4. caffeine intake 100-400 mg/d; and
5. ability to participate in physical activity for a minimum of 150 min/week.

Exclusion Criteria:

1. pregnancy, lactation or actively trying to become pregnant;
2. medical illnesses or medications that could affect body weight;
3. cigarette smokers;
4. weight loss of 10 or more pounds in the last 3 months;
5. fasting blood glucose greater than 126mg/dl;
6. participation in a clinical research study that would conflict with the purpose of the current trial; and
7. other factors that in the judgment of the principal investigator may interfere with study participation or the ability to follow the intervention protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
body weight | 12 weeks
  Body weight is assessed at baseline, 6 and 12 weeks. Body weight is determined using a calibrated scale.

SECONDARY OUTCOMES:
DEXA-determined fat mass | 12 weeks
  Body fat percent is determined by DEXA using a whole body scanner.

CONTACTS AND LOCATIONS:
Overall Officials: John P Foreyt, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (2):
  - Temple University, Philadelphia, Pennsylvania
  - Behavioral Medicine Research Center, Houston, Texas
- MRC Human Nutrition Research, Cambridge, United Kingdom